CLINICAL TRIAL: NCT01900132
Title: Electrical Impedance Myography: Natural History Studies in Neuromuscular Disorders and Healthy Volunteers
Brief Title: Electrical Impedance Myography: Natural History Studies inNeuromuscular Disorders and Healthy Volunteers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 130165; 13-N-0165
Record Dates: First submitted 2013-07-11; First posted 2013-07-16 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-05-15

CONDITIONS: Neuromuscular Disease; Motor Neuron Disease; Inherited Neuromuscular Conditions; Inherited Neuropathies
Keywords: Electrophysiology; Neuromuscular Disease
MeSH Terms: conditions — Neuromuscular Diseases; Motor Neuron Disease | interventions — Nerve Conduction Studies; Electromyography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1/All Subjects (Experimental): Healthy Volunteers and patients
  Interventions: Device: EIM testing; Device: Nerve & muscle ultrasonography; Device: Nerve conduction studies; Device: Electromyography (EMG)

INTERVENTIONS:
Device: EIM testing — EIM device is placed on the muscle and a high frequency current is delivered to the skin.
Device: Nerve & muscle ultrasonography — Ultrasound waves to examine the muscles and nerves
Device: Nerve conduction studies — Small metal disk electrodes attached to wires onto skin to measure how fast nerves conduct electrical impulses and the strength of the connection between nerves and muscles.
Device: Electromyography (EMG) — Thin needle placed into muscles to record electrical activity-adults only

SUMMARY:
Background:

- Electrical impedance myography (EIM) is a new technique being studied to see if it is helpful in evaluating muscle disorders and nerve disorders. EIM looks at how a mild, painless electrical current travels through muscles. Researchers want to gain experience in using the EIM device. They will collect information on the results of using it on people with and without nerve and muscle diseases, and compare that with information from other standard tests. First, they will test the device on healthy people. Then they will test people with a variety of neuromuscular diseases. Because the test is noninvasive and not painful, researchers will test both children and adults.

Objectives:

- To gain experience using the EIM muscle testing device.

Eligibility:

* Healthy volunteers at least 2 years old.
* Individuals at least 2 years old who have neuromuscular disease.

Design:

* Participants will be screened with a medical history and physical exam.
* Participants will have one 2-3 hour clinic visit. Researchers may request follow-up visits.
* Participants will be tested with the EIM device. The device and small electrodes will be placed on their skin. An electric current will pass through the device, but the participants will not feel this.
* Participants may have an ultrasound test. A gel will be put on their skin, and a device will be moved over the skin.
* Participants may have a nerve test. Electrodes will be placed on their skin, and they will feel a small shock.
* Participants may have a test where a thin needle is inserted in their muscle.

DETAILED DESCRIPTION:
Title: Electrical Impedance Myography: Natural History Studies in Neuromuscular Disorders and Healthy Volunteers

Study Description: This is a natural history study examining the utility of electrical impedance myography (EIM) device in the evaluation of neuromuscular disorders. This is a novel device so the initial step was to establish reproducibility of the data and expected normative values using the EIM device on healthy volunteers. In neuromuscular disorders, the EIM device will be used to understand the results in different types of neuromuscular disorders. A subset of subjects with neuromuscular disorders are studied serially as preliminary evaluation of its utility as a biomarker in clinical studies. The protocol includes both adult and pediatric subjects.

Objectives:

Primary objective: For subjects with neuromuscular disease, we aim to understand if EIM has utility in differentiating neuromuscular disorders in adult and pediatric subjects. Also, to perform preliminary serial studies to understand the EIM device potential use as biomarker in clinical studies.

For healthy volunteers, the primary objective is reproducibility of results and the range of normative values in adult and pediatric subjects.

Secondary objectives: The three parameters, phase, reactance, resistance will be followed serially as measures of change in pediatric population.

As exploratory outcome measures, we will explore correlations between EIM and ultrasound and other electrodiagnostic methods.

Endpoints:

Primary endpoint:

For healthy volunteers, intra and interrater reliability will be evaluated to determine the utility of EIM as a reproducible biomarker. Normative values will be developed using a range of ages, mixed gender, and race to be used as a basis of comparison with subjects with neuromuscular disorders.

For subjects with neuromuscular disorders, patterns of phase, resistance and reactance in different types of neuromuscular disorders will be evaluated and examined for patterns specific to type of neuromuscular disorder.

Secondary endpoint:

The three parameters, phase, reactance, resistance will be followed serially as measures of change. This will be in evaluated small groups of neuromuscular disorders that are referred to this protocol. A cohort of pediatric healthy volunteers will be followed for two years for comparative data with pediatric subjects with neuromuscular disorders.

Exploratory endpoint:

The EIM phase, muscle ultrasound and possibly MUNIX will be compared in healthy volunteers.

Study Population: 275

(150) Patients with neuromuscular disease, over age 2

(125) Healthy Volunteers; 90 adults age 18 and above; 35 children age 7 to 17.

Description of Sites/Facilities Enrolling Participants:All studies will be performed in the NIH Clinical Center. The majority of the studies will occur in the EMG Lab. The EMG Lab is an AANEM-accredited EMG lab to perform diagnostic electrodiagnostic studies with experience in both pediatric and adult populations. At the convenience for the subject, the EIM study can be performed in other parts of the NIH Clinical Center.

Study Duration: It is estimated that the duration of the study will be 10 years. With closure in 2023.

Participant Duration: For the healthy volunteers, we will be evaluating EIM along with possible ultrasound and electrodiagnostic methods. A single session will be 3 hours or less. Repeat studies may be performed to establish reproducibility after the initial studies are completed. For subjects with neuromuscular disease, the studies will be conducted in a single outpatient session of 3 hours or less, unless a follow-up study is requested by the primary team. For children, the session will be 2 hours or less.

ELIGIBILITY:
* INCLUSION CRITERIA:

HEALTHY VOLUNTEERS-ADULTS

1. Healthy adults, male or female, aged 18 years old or older,
2. In good general health as evidenced by medical history
3. Stated willingness to comply with all study procedures and availability for the duration of the study.
4. Ability of subject to understand and the willingness to sign a written informed consent document.

HEALTHY VOLUNTEERS-PEDIATRIC

1. Healthy children, male or female, age 7-18,
2. In good general health as evidenced by medical history
3. Stated willingness to comply with all study procedures and availability for the duration of the study
4. Ability of subject or Legally Authorized Representative (LAR)) to understand and the willingness to sign a written informed consent document.

SUBJECTS WITH NEUROMUSCULAR DISEASE

Adult and pediatric, male or female, patients with a neuromuscular disorder are eligible even if the exact etiology of the disorder is unknown at the time of enrollment into this study. This will include neuropathy, myopathy and motor neuron disorders. It is expected that the subjects are undergoing appropriate standard diagnostic and genetic work-up outside of this protocol that will later clarify the specific etiology of the disorder. Movement disorder will also be included because of the prior research done on dystonia and EIM.

Inclusion criteria

1. Suspected motor neuron disease or
2. Suspected myopathy or
3. Suspected neuropathy or
4. Suspected movement disorders that impair intracortical processes
5. Age of 2 years or older
6. Ability of subject to sign a written informed consent document.

NIH EMPLOYEES:

NIH employees and staff may participate, however EMG Section, OCD, NINDS, employees may not participate.

EXCLUSION CRITERIA:

HEALTHY VOLUNTEERS-ADULTS

1. Medical conditions that require medications that affects the physiological measures being tested. Some conditions that may be excluded are diabetes, kidney and liver disease.
2. History of stroke, muscle disorders, peripheral neuropathy or spine surgery

HEALTHY VOLUNTEERS-PEDIATRIC

1. Medical conditions that require medications that affects the physiological measures being tested. Some conditions that may be excluded are diabetes, kidney and liver disease.
2. History of stroke, muscle disorders, peripheral neuropathy or spine surgery

SUBJECTS WITH NEUROMUSCULAR DISEASE:

No clinical evidence of a neuromuscular disorder on clinical evaluation.

Ages: 2 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2013-06-20 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Patients - EIM measures for a selection of muscles | End of study
  Obtaining measures using EIM device in different types of neuromuscular disorders.
Healthy Volunteers - EIM measures for a selection of muscles with the aim of developing normative values for the NIH EMG lab | End of study
  Obtaining measures using EIM device- reproducibility and normative data

SECONDARY OUTCOMES:
Serial studies in pediatric patients | End of study
  Serial measures of EIM in patients with neuromuscular disorders
Healthy Volunteers - exploratory correlations of ultrasound and electrodiagnostic methods such nerve conduction studies and less likely, EMG | End of study
  Obtaining measures using EIM device and comparing with ultrasound and motor unit number estimation techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya J Lehky, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
There is no formalized plan to make IPD available of a website. The data from this protocol would be available in anonomyzed format in relationship to publications.

REFERENCES:
- [Background] Nichols C, Jain MS, Meilleur KG, Wu T, Collins J, Waite MR, Dastgir J, Salman A, Donkervoort S, Duong T, Keller K, Leach ME, Lott DJ, McGuire MN, Nelson L, Rutkowski A, Vuillerot C, Bonnemann CG, Lehky TJ. Electrical impedance myography in individuals with collagen 6 and laminin alpha-2 congenital muscular dystrophy: a cross-sectional and 2-year analysis. Muscle Nerve. 2018 Jan;57(1):54-60. doi: 10.1002/mus.25629. Epub 2017 Apr 25. PMID 28224647
- [Background] Schwartz DP, Dastgir J, Salman A, Lear B, Bonnemann CG, Lehky TJ. Electrical impedance myography discriminates congenital muscular dystrophy from controls. Muscle Nerve. 2016 Mar;53(3):402-6. doi: 10.1002/mus.24770. Epub 2015 Aug 13. PMID 26179210
- [Background] Offit MB, Wu T, Floeter MK, Lehky TJ. Electrical impedance myography (EIM) in a natural history study of C9ORF72 mutation carriers. Amyotroph Lateral Scler Frontotemporal Degener. 2020 Aug;21(5-6):445-451. doi: 10.1080/21678421.2020.1752247. Epub 2020 Apr 21. PMID 32312103
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-N-0165.html